CLINICAL TRIAL: NCT04807569
Title: A Prospective Randomized Trial "The Effectiveness of Peripheral Magnetic Stimulation in Men With Lower Urinary Tract Symptoms"
Brief Title: The Effectiveness of Peripheral Magnetic Stimulation in Men With Lower Urinary Tract Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Joint-Stock Company North-West Center for Evidence-Based Medicine, Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2/2021
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Bladder Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 10 sessions of non-invasive peripheral magnetic neuromodulation using the BTL Emsella magnetic stimulator according to the manufacturer's standard protocol: "pelvic floor rehabilitation".
  Interventions: Other: Peripheral magnetic neuromodulation
- Control group (Experimental): one-month course of drug therapy with alpha-1-adrenoblocker according to the standard scheme
  Interventions: Drug: Taking drug Tamsulosin

INTERVENTIONS:
Other: Peripheral magnetic neuromodulation — Non-invasive peripheral magnetic neuromodulation using the BTL Emsella magnetic stimulator according to the manufacturer's standard protocol: "pelvic floor rehabilitation
  Arms: Experimental group
Drug: Taking drug Tamsulosin — Tamsulosin at a dose of 0.4 mg x 1 time per day orally for 1 month.
  Arms: Control group

SUMMARY:
The main hypothesis of this study is that peripheral magnetic neuromodulation can correct the symptoms of lower urinary tract in men. We assume that under the influence of t peripheral magnetic stimulation, both the subjective state of patients assessed by standardized questionnaires and a urination diary, as well as the objective parameters, assessed by non-invasive urodynamic studies, will be improved. This study will use standard protocols built into the BTL Emsella magnetic stimulator.

DETAILED DESCRIPTION:
The aim of the study is to test the hypothesis that the use of the peripheral magnetic stimulation in men with lower urinary tract symptoms will help to reduce subjective and objective clinical symptoms and improve the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Signed informed consent;
3. The presence of lower urinary tract symptoms: urinary frequency, nocturia, urgency; feeling of incomplete bladder, weak urine stream.

Exclusion Criteria:

1. The patient, who have been implanted devices that control physiological functions (a pacemaker, a device for deep brain stimulation and chronic epidural brain stimulation, a cochlear implant).
2. Convulsive attacks in the anamnesis;
3. Taking medications that may trigger the risk of seizures;
4. The presence in the patient's body of metal elements or objects made with the use of ferromagnets (joint prostheses, eye prostheses, tattoos made using metal ink, surgical clips, staples and other metal suture materials, etc.)
5. Chronic cardiovascular and cerebrovascular diseases in the stage of decompensation or recent acute conditions (myocardial infarction, brain stroke, etc.)
6. The presence of infravesical obstruction in men, determined by uroflowmetry (obstructive urination curve according to the Liverpool nomogram);
7. The postvoid residual volume (more than 50 ml);
8. The concentration of prostate specific antigen (PSA) in the blood is more than 4.0 ng / ml;
9. The presence of urinary tract infection;
10. A history of cancer of the pelvic floor organs;

Ages: 25 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
IPSS change score | Baseline, 4, 12, 24, 48 weeks
  The IPSS questionnaire evaluates the impact of lower urinary tract symptoms on the patient's quality of life. It consists of 8 questions. Questionts evaluates whether the patient has symptoms of incomplete emptying of the bladder and ranges from 0 to 5 points. The increase in scores is directly proportional to the increase in symptoms.
Change baseline of micturition episodes per day | Baseline, 4, 12, 24, 48 weeks
  Patients should document how many times they go to the restroom during the day and at night, as well as the loss of urine in stressful situations (coughing, sneezing, laughter, squatting, weightlifting, walking, running), changing liner or absorbent and episodes of urgency and urgency-incontinence. The journal shall be held for a consecutive period of 24 hours, for a minimum of three consecutive days.

SECONDARY OUTCOMES:
Change baseline of micturition episodes per day | Baseline, 4, 12, 24, 48 weeks
  Patients should document how many times they go to the restroom during the day and at night, as well as the loss of urine in stressful situations (coughing, sneezing, laughter, squatting, weightlifting, walking, running), changing liner or absorbent and episodes of urgency and urgency-incontinence. The journal shall be held for a consecutive period of 24 hours, for a minimum of three consecutive days.

CONTACTS AND LOCATIONS:
Locations (1):
- Joint-Stock Company "North-Western Centre of Evidence-Based Medicine", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No